CLINICAL TRIAL: NCT04432688
Title: The Safety and Effectiveness of Latuda® Post-marketing Surveillance in the Treatment of Chinese Schizophrenia Patients
Status: Completed | Type: Observational
Sponsor: Sumitomo Pharma (Suzhou) Co., Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: DSPCLAT-001
Record Dates: First submitted 2020-06-09; First posted 2020-06-16 (Actual); Last update posted 2024-04-18 (Actual); Status verified 2024-04

CONDITIONS: Schizophrenia
MeSH Terms: conditions — Schizophrenia | interventions — Lurasidone Hydrochloride

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Weeks
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

GROUPS / COHORTS (1):
- Latuda®: Chinese schizophrenia patients who are receiving Latuda® in the real world
  Interventions: Drug: Lurasidone HCl

INTERVENTIONS:
Drug: Lurasidone HCl — This is a non-interventional, observational study
  Other Names: Latuda®

SUMMARY:
It's a prospective, non-interventional, observational Post-marketing Surveillance..

DETAILED DESCRIPTION:
It's a prospective, non-interventional, observational Post-marketing Surveillance, the aim of the surveillance is to observe the safety and overall effectiveness of Latuda® in the treatment of Chinese patients with schizophrenia for 12 weeks in real clinical practice, as well as the dose of Latuda® for monotherapy or combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* Schizophrenia Patients who begin to receive Latuda®

Exclusion criteria:

* No exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Schizophrenia Patients who begin to receive Latuda®
Sampling Method: Non-Probability Sample
Enrollment: 3192 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2023-03-18 (Actual); Study Completion 2023-06-18 (Actual)

PRIMARY OUTCOMES:
The incidence of Adverse Event | week 12
  Adverse events

SECONDARY OUTCOMES:
The incidence of extrapyramidal symptom | baseline/ week 2-4/ week 6-8/ week 12
  Extrapyramidal Symptoms (EPS) are drug-induced movement disorders that accur due to antipsychotic blockade of the nigrostriatal dopamine tracts, including acute dystonia, akathisia, antipsychotic-induced parkinsonism, tardive dyskinesia (TD)
The incidence of akathisia | baseline/ week 2-4/ week 6-8/ week 12
  Akathisia is a side effect of antipsychotic drugs, presenting as restlessness, fidgeting of the legs, rocking, pacing, and the inability to sit or stand still.
the rate of use of extrapyramidal symptom treatment drugs | baseline/ week 2-4/ week 6-8/ week 12
  extrapyramidal symptom treatment drugs are medications to decrease extrapyramidal side effects
Changes in body weight at the end of treatment compared with baseline | baseline/ week 12
  Weight is measured on a scale
The overall Brief Psychiatric Rating Scale (BPRS) score change at the end of the treatment compared with the baseline | baseline/ week 2-4/ week 6-8/ week 12
  Brief Psychiatric Rating Scale (BPRS) is a generic scale developed to measure clinical change in patients with schizophrenia and which can be used as a global measure of psychopathology. Each of the 18 items are designed to represent a discrete symptom area. Items are rated on a 7-point Likert scale, from 1 = "not present" to 7 = "extremely severe", with scores ranging from 18 to 126 (achieved through summing the item scores).

CONTACTS AND LOCATIONS:
Overall Officials: Yifeng Xu, Principal Investigator — Shanghai Mental Health Center
Locations (7):
- China (7):
  - Beijing Anding Hospital, Beijing, Beijing Municipality
  - The first specialized hospital of Harbin, Harbin, Heilongjiang
  - Brain Hospital of Hunan Province, Changsha, Hunan
  - Shandong Mental Health Center, Jinan, Shandong
  - Shanghai Mental Health Center, Shanghai, Shanghai Municipality
  - First Affiliated Hospital of Shanxi Medical University, Taiyuan, Shanxi
  - Tianjin Anding Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No